CLINICAL TRIAL: NCT03010319
Title: Prospective, Multi-center, Randomized, Controlled Trial Evaluating the Use of PriMatrix Dermal Repair Scaffold for the Management of Diabetic Foot Ulcers
Brief Title: PriMatrix for the Management of Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T-PMXDFU-001
Record Dates: First submitted 2017-01-03; First posted 2017-01-05 (Estimated); Results first posted 2022-03-15 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PriMatrix (Experimental): Arm will receive PriMatrix Dermal Repair Scaffold plus secondary dressings to maintain a moist wound healing environment and an appropriate off-loading device.
  Interventions: Device: PriMatrix Dermal Repair Scaffold; Device: Secondary Dressings; Device: Offloading device
- Standard of Care (Active Comparator): Arm will receive moist wound therapy consisting of 0.9% Sodium Chloride gel plus secondary dressings and an appropriate off-loading device.
  Interventions: Device: Secondary Dressings; Device: Offloading device

INTERVENTIONS:
Device: PriMatrix Dermal Repair Scaffold — Application of PriMatrix to ulcer
  Arms: PriMatrix
Device: Secondary Dressings — Dressings to ensure moist wound environment
Device: Offloading device — Offloading device to decrease pressure to wound area

SUMMARY:
The study will evaluate the efficacy of PriMatrix Dermal Repair Scaffold in the management of diabetic foot ulcers in subjects with diabetes mellitus versus the Standard of Care treatment. Half of patients will be treated using PriMatrix while the other half will receive Standard of Care treatment.

DETAILED DESCRIPTION:
A diabetic foot ulcer (DFU) is a major health complication that affects up to 15% of individuals with diabetes mellitus over their lifetime. The treatment of DFUs is extremely challenging as these ulcers may not respond to standard of care (SC) treatment and frequently become infected.

Advanced wound therapies like PriMatrix have become an important strategy in the treatment of hard-to-heal chronic DFUs by trapping and binding the patients' own cells to rebuild the dermis layer of the skin to aid in healing.

The study will evaluate the efficacy of PriMatrix Dermal Repair Scaffold in the closure of DFUs in subjects with diabetes mellitus in comparison to Standard of Care treatment.

ELIGIBILITY:
Inclusion Criteria

Subjects are required to meet all of the following criteria for enrollment into the study and subsequent randomization:

1. The subject has signed and dated an informed consent form.
2. In the opinion of the investigator, subject is able and willing to comply with study procedures, including study visits, study dressing regimens and compliance with study required off-loading device.
3. The subject is ≥ 18 years of age.
4. The subject, if female of child-bearing potential, must not be pregnant. To document pregnancy status, subject statement is acceptable.
5. The subject has Type I or Type II diabetes mellitus with investigator-confirmed glycosylated hemoglobin (HbA1c) of ≤ 12% within 3 months prior to screening visit.
6. The subject has at least one diabetic foot ulcer that meets ALL of the following criteria:

   * Ulcer which has been in existence for a minimum of two weeks, prior to signing the Informed Consent Form for trial participation.
   * Ulcer is a partial or full thickness diabetic foot ulcer without capsule/tendon/bone exposure.
   * Ulcer does not have tunneling, undermining, or sinus tracts that necessitates surgical OR debridement and/or penetrates to capsule/tendon/bone.
   * Ulcer is located on the foot or ankle (with no portion above the top of the malleolus).
   * Ulcer size (area) is > 1 cm2 and < 12 cm2 post-debridement.
7. There is a minimum 1 cm margin between the qualifying study ulcer and any other ulcer on that same foot, post-debridement.

   • If the subject has more than one ulcer that meets the eligibility criteria, the ulcer designated as the study ulcer will be at the discretion of the investigator.
8. The subject has adequate vascular perfusion of the affected limb as defined by at least one of the following:

   * Ankle-Brachial Index (ABI) ≥ 0.65 or ≤1.2, performed within 3 months of screening,
   * Toe pressure (plethysmography) > 50 mmHg at time of screening,
   * TcPO2 > 40 mmHg at time of screening
9. The subject or responsible caregiver is willing and able to maintain required applicable dressing changes as well as study required off-loading/protective device for the duration of the study.

Exclusion Criteria

Subjects will not be enrolled in the study if any of the following criteria are met:

1. The subject was previously randomized and treated under this clinical study protocol.
2. The subject has suspected or confirmed gangrene or ulcer infection of the study ulcer or receiving systemic antibiotics for the treatment of such.
3. The subject has suspected or confirmed osteomyelitis of the foot with the study ulcer.
4. The subject has a history of hypersensitivity to bovine collagen, as determined by prior medical history.

   Protocol Number: T-PMXDFU-01 Confidential Page 23 of 64 Version 5.0 06 Nov 2018
5. The subject has participated in another clinical trial involving a device or a systemically administered investigational study drug/treatment within 28 days of randomization.
6. The subject has received, within 28 of signing Informed Consent Form, or is scheduled to receive during study participation, a medication or treatment which is known to interfere with or affect the rate and quality of ulcer healing (e.g., systemic steroids, immunosuppressive therapy, autoimmune disease therapy, dialysis, radiation therapy to the foot, vascular surgery, angioplasty, or thrombolysis).
7. The subject has a history of bone cancer or metastatic disease of the affected limb, radiation therapy to the foot, or has had chemotherapy within the 12 months prior to signing Informed Consent Form for trial participation.
8. In the opinion of the investigator, the subject has a history of, or is currently diagnosed with, any illness or condition, other than diabetes, that could interfere with ulcer healing (e.g., end-stage renal disease, severe malnutrition, liver disease, aplastic anemia, connective tissue disorder, acquired immune deficiency syndrome, HIV positive, or sickle cell anemia).
9. In the opinion of the investigator, the subject has unstable Charcot foot or Charcot with bony prominence that could inhibit ulcer healing.
10. The subject has ulcers secondary to a disease other than diabetes (e.g., vasculitis, neoplasms, or hematological disorders).
11. In the opinion of the investigator, the subject has excessive lymphedema that could interfere with off-loading and/or ulcer healing.
12. The study ulcer has received ulcer dressings that included growth factors, engineered tissues, or skin substitutes within 28 days of randomization or is scheduled to receive treatment during the study (e.g., Regranex, Dermagraft, Apligraf, EpiFix, GraftJacket, OASIS, Omnigraft, or Integra BMWD).
13. At the end of the screening phase and based on planimetric assessment, the area of the study ulcer after sharp debridement has decreased by more than 30% over the two-week screening period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Lantis, MD, Principal Investigator — The Mount Sinai Medical Center
Locations (17):
- United States (17):
  - ILD Research Center, Carlsbad, California
  - LA Foot & Ankle Clinic, Los Angeles, California
  - Center for Clinical Research, Inc., San Francisco, California
  - Central Valley Vein and Wound, Selma, California
  - Georgetown University, Washington D.C., District of Columbia
  - Barry University Clinical Research, North Miami, Florida
  - LA Podiatry Group, West Palm Beach, Florida
  - Podiatry 1st, Belleville, Illinois
  - The Mount Sinai Medical Center, New York, New York
  - Wound Care of Tulsa, Tulsa, Oklahoma
  - Martin Foot and Ankle, York, Pennsylvania
  - Podiatric Medical Partners of Texas, P.A., Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - JPS Health Network, Fort Worth, Texas
  - Futuro Clinical Trials, McAllen, Texas
  - Element Research Group, San Antonio, Texas
  - Foot and Ankle Institute, St. George, Utah

IPD SHARING:
Plan to Share IPD: No
Individual Patient Data will not be shared.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PriMatrix | Standard of Care
Started | 110 | 116
Completed | 84 | 87
Not Completed | 26 | 29
Not completed — Adverse Event | 15 | 9
Not completed — Withdrawal by Subject | 1 | 6
Not completed — Physician Decision | 2 | 4
Not completed — Sponsor requested withdrawal | 2 | 2
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Other Reason | 5 | 7

BASELINE CHARACTERISTICS:
Population: Primary Efficacy Population
Groups:
- Total: Total of all reporting groups
Arm/Group | PriMatrix | Standard of Care | Total
Number analyzed (Participants) | 103 | 104 | 207
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.5 (11.92) | 57.6 (11.49) | 58.0 (11.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 24 | 44
  Male | 83 | 80 | 163
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 43 | 31 | 74
  Not Hispanic or Latino | 60 | 73 | 133
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 19 | 26 | 45
  White | 81 | 74 | 155
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 103 | 104 | 207

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Complete Wound Closure, as Assessed by the Investigator, at or Before Week 12 of the Treatment Phase
Description: Complete wound closure was defined as 100% re-epithelialization of the ulcer surface without detectable exudate, confirmed on 2 consecutive study visits 1 week apart.
Time Frame: 12-week Treatment Phase
Population: Primary Efficacy Population
Measure: Count of Participants; unit: Participants
Arm/Group | PriMatrix | Standard of Care
Number analyzed (Participants) | 103 | 104
Participants | 47 | 29

2. Secondary Outcome: Percentage of Subjects With Complete Wound Closure, as Assessed by Computerized Planimetry, at or Before Week 12 of the Treatment Phase
Time Frame: 12-week treatment phase
Population: Primary Efficacy Population
Measure: Count of Participants; unit: Participants
Arm/Group | PriMatrix | Standard of Care
Number analyzed (Participants) | 103 | 104
Participants | 36 | 20

3. Secondary Outcome: Time to Complete Wound Closure, as Assessed by the Investigator
Time Frame: 12-week Treatment Phase
Population: Primary Efficacy Population with Complete Wound Closure
Measure: Mean (Standard Deviation); unit: days
Arm/Group | PriMatrix | Standard of Care
Number analyzed (Participants) | 47 | 29
days | 53.6 (21.39) | 56.2 (18.24)

4. Secondary Outcome: Time to Complete Wound Closure, as Assessed by Computerized Planimetry.
Time Frame: 12-week Treatment Phase
Population: Primary Efficacy Population with Complete Wound Closure
Measure: Mean (Standard Deviation); unit: days
Arm/Group | PriMatrix | Standard of Care
Number analyzed (Participants) | 36 | 20
days | 51.8 (20.63) | 56.8 (16.25)

5. Secondary Outcome: Rate of Wound Closure, as Assessed by Computerized Planimetry.
Description: Rate of Wound closure was recorded as the percentage of the wound that was closed, per week.
  NOTE1: Rate (% closed/week) = 7 * [(Baseline wound size) - (Post-baseline wound size)]/[(Baseline wound size) * (days in trial)] NOTE2: Missing data is imputed using LOCF method for this analysis
Time Frame: Weeks 1-12 during Treatment Phase
Population: Primary Efficacy Population
Measure: Mean (Standard Deviation); unit: Percentage of Wound Closed/Week
Arm/Group | PriMatrix | Standard of Care
Number analyzed (Participants) | 103 | 104
Percentage of Wound Closed/Week
  Week 1 | 1.727 (7.142) | 0.996 (8.222)
  Week 2 | 1.722 (9.446) | 1.999 (9.366)
  Week 3 | 2.587 (10.082) | 2.524 (9.304)
  Week 4 | 3.443 (9.376) | 2.990 (9.653)
  Week 5 | 3.603 (9.371) | 3.476 (9.549)
  Week 6 | 3.764 (9.441) | 3.279 (9.951)
  Week 7 | 4.054 (9.402) | 3.308 (10.072)
  Week 8 | 4.017 (9.759) | 3.632 (10.115)
  Week 9 | 4.213 (9.554) | 3.820 (10.184)
  Week 10 | 3.970 (10.230) | 3.896 (10.184)
  Week 11 | 4.558 (9.480) | 3.837 (10.186)
  Week 12 | 4.637 (9.513) | 3.928 (10.263)

ADVERSE EVENTS:
Time Frame: Adverse Events data was collected from Screening Visit 2 through a potential Four-Week Post Wound Closure Visit, for a total of up to 17 weeks.
Description: Adverse Event Reporting population is the Safety Population.
Arm/Group | PriMatrix | Standard of Care
All-Cause Mortality (participants affected / at risk) | 1/110 | 0/116
Serious Adverse Events (participants affected / at risk) | 19/110 | 15/116
Other Adverse Events (participants affected / at risk) | 16/110 | 23/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PriMatrix (N=110) | Standard of Care (N=116)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Catheter site thrombosis (General disorders) | 1 (1) | 0 (0)
Chest Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 2 (2)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
Diabetic foot infection (Infections and infestations) | 3 (3) | 7 (7)
Gangrene (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 8 (8) | 3 (3)
Septic Shock (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary Track Infection (Infections and infestations) | 1 (1) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Shock hypoglycemic (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Coronary artery bypass (Surgical and medical procedures) | 1 (1) | 0 (0)
Foot amputation (Surgical and medical procedures) | 0 (0) | 1 (1)
Metatarsal excision (Surgical and medical procedures) | 1 (1) | 0 (0)
Angiopathy (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Peripheral ischemia (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PriMatrix (N=110) | Standard of Care (N=116)
Diabetic Foot Infection (Infections and infestations) | 8 (8) | 11 (11)
Diabetic Foot (Infections and infestations) | 8 (8) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators are barred from publishing or disclosing results until a multicenter publication is published or until a period of 24 months after study completion passes, whichever comes first.

DOCUMENTS (2):
  • Study Protocol (2018-11-06): https://cdn.clinicaltrials.gov/large-docs/19/NCT03010319/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-19): https://cdn.clinicaltrials.gov/large-docs/19/NCT03010319/SAP_001.pdf